CLINICAL TRIAL: NCT06809270
Title: Liver Function and Inflammation in Obese Postmenopausal Women: Responses to Moderate Intensity Intermittent Walking
Brief Title: Moderate Intensity Intermittent Walking in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wissal Abassi (Other)
Responsible Party: Sponsor-Investigator, Wissal Abassi, Principal Investigator, High Institute of Sports and Physical Education of Kef
Organization: High Institute of Sports and Physical Education of Kef (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Walking and liver function
Record Dates: First submitted 2025-01-25; First posted 2025-02-05 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-01

CONDITIONS: Liver Enzymes; Inflammatory Markers
Keywords: Alanine transaminase; Alkaline phosphatase; Postmenopausal obesity; C-reactive protein; Walking training; Erythrocyte sedimentation rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): The training group underwent a moderate intensity intermittent walking training at 60% to 80% of the 6-min-walking-test distance, four times a week of 60 min/session for a period of 10 weeks.
  Interventions: Behavioral: Walking training intervention
- Control group (No Intervention): No training intervention was intended for this group.

INTERVENTIONS:
Behavioral: Walking training intervention — Moderate intensity intermittent walking training for a period of 10 weeks. The intensity of the training is 60 to 80% of 6MWTdistance. The frequency of the training is four times a week.
  Arms: Training group

SUMMARY:
The goal of this clinical trial is to investigate the impact of a walking training intervention program on liver enzymes and selected inflammatory markers in postmenopausal women with obesity. The main question it aims to answer is:

Does walking training reduce the risk of liver disease by modulating hepatic-enzymes and selected inflammatory markers? Researchers will compare walking training intervention (designed to the experimental group) to non-training intervention (designed to the control group) to see if the training program works to improve liver health in obese postmenopausal women.

Participants in the experimental (training) group will: underwent a moderate intensity intermittent walking training (MIWT) at 60% to 80% of the 6-min-walking-test distance, four times a week of 60 min/session.

Participants in control group will : not perform any physical training and maintain their usual daily activities.

DETAILED DESCRIPTION:
Postmenopausal obesity is an important public health problem accompanied by increased systemic inflammation that escalates the risk of liver disease. Exercise improved inflammatory and hepatic function. Moderate-intensity intermittent-walking-training (MIWT) is the most feasible for obese-postmenopausal-women. This study aimed to investigate whether MIWT could reduce the risk by modulating hepatic-enzymes and selected inflammatory markers. Thirty-six sedentary obese postmenopausal women (mean age 55.7±3.5) were randomly divided into two groups: training group (TG, n=18) and control group (CG, n=18). The TG underwent a MIWT at 60% to 80% of the 6-min-walking-test distance, four times a week of 60 min/session. Body composition, hepatic (alanine-transaminase (ALT), aspartate-transaminase (AST), alkaline-phosphatase, gamma-glutamyl-transferase (GGT) and serum-bilirubin] and inflammatory markers [C-reactive-protein (CRP), and erythrocyte-sedimentation-rate (ESR)) were evaluated at baseline and after 10-week of protocol.

ELIGIBILITY:
Inclusion Criteria:

Women included are:

* Postmenopausal (≥1 year of amenorrhea).
* Obese (body mass index (BMI) ≥30 kg/m2).
* Sedentary (<120 min/week of low to moderate intensity physical activity at during the past 6 months).
* Aged 50 to 60 years.

Exclusion Criteria:

* Suffering from any cardiovascular/renal/pulmonary/metabolic disease.
* Being under menopausal hormone therapy.
* Presenting any orthopedic limitations interfering the ability to perform the study intervention.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2024-12-22 (Actual); Study Completion 2024-12-22 (Actual)

PRIMARY OUTCOMES:
Alanine transaminase | At baseline and at week 11(after the ten weeks of the training intervention).
  Serum concentrations of alanine-transaminase (ALT) are measured from a blood sample (5 ml) using a Chemistry System Analyzer (Beckman Coulter AU480, France).
Aspartate transaminase | At baseline and at week 11(after the ten weeks of the training intervention).
  Serum concentrations of aspartate-transaminase (AST),are measured from a blood sample (5 ml) using a Chemistry System Analyzer (Beckman Coulter AU480, France).
Alkaline phosphatase | At baseline and at week 11(after the ten weeks of the training intervention).
  Serum concentrations of alkaline-phosphatase are measured from a blood sample (5 ml) using a Chemistry System Analyzer (Beckman Coulter AU480, France).
Gamma glutamyl transferase | At baseline and at week 11(after the ten weeks of the training intervention)
  Serum concentrations of gamma-glutamyl-transferase (GGT),are measured from a blood sample (5 ml) using a Chemistry System Analyzer (Beckman Coulter AU480, France).
Serum bilirubin | At baseline and at week 11(after the ten weeks of the training intervention).
  Serum concentrations of bilirubin are measured from a blood sample (5 ml) using a Chemistry System Analyzer (Beckman Coulter AU480, France).
C reactive protein | At baseline and at week 11(after the ten weeks of the training intervention).
  Serum concentration of C-reactive-protein (CRP) are measured from a blood sample (5 ml).
Erythrocyte sedimentation rate | At baseline and at week 11(after the ten weeks of the training intervention).
  Erythrocyte-sedimentation-rate (ESR) are measured from a blood sample (5 ml).

SECONDARY OUTCOMES:
Body composition | At baseline and after ten weeks of the training intervention.
  Body composition were determined, with barefoot and lightly dressed subjects, using a stadiometer (Holtain Ltd., UK) and an electronic scale (Tanita BC-533, Tokyo, Japan).
Aerobic capacity | At baseline and after ten weeks of the training intervention.
  The 6-minute walk test was performed before and after the training intervention as an indicator of exercise capacity.

CONTACTS AND LOCATIONS:
Locations (1):
- High Institute of Sports and Physical Education of Kef, Boulifa, Kef Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No
For confidentiality reasons, all data from this study are available upon request.